CLINICAL TRIAL: NCT04490889
Title: Noninvasive Preimplantation Genetic Testing for Aneuploidy Using Cell Free DNA on Spent Culture Media
Brief Title: Noninvasive Preimplantation Genetic Testing for Aneuploidy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mỹ Đức Hospital (Other)
Collaborators: My Duc Phu Nhuan Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: CS/BVMĐ/20/11
Record Dates: First submitted 2020-07-24; First posted 2020-07-29 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Preimplantation Genetic Testing (PGT); ICSI
Keywords: NiPGT-A; Cell free DNA (cfDNA); SCM; Sensitivity
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — TE biopsy of blastocyst and cfDNA into spent culture media.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with PGT indication: Patients undergo in vitro fertilization with PGT-A or for PGT-SR indication
  Interventions: Diagnostic Test: NiPGT-A

INTERVENTIONS:
Diagnostic Test: NiPGT-A — NiPGT-A is the technique to screen the aneuploidy status of an embryo without invasion technique, such as biopsy. We use SCM to isolate cfDNA, then amplify and analyse the aneuploidy of embryo secreting this material using NGS technique.

SUMMARY:
The study is conducted to evaluate the sensitivity and specificity of non-invasive preimplantation genetic testing for aneuploidy (NiPGT-A) using cell free DNA into spent culture medium (SCM).

DETAILED DESCRIPTION:
Our study is a diagnostic study, recruit 218 biopsied blastocysts from couples undergoing intracytoplasmic sperm injection (ICSI) with Preimplantation genetic testing for aneuploidy (PGT-A) or Preimplantation genetic testing for structural rearrangements (PGT-SR) indication.

Oocyte retrieval, ICSI and embryo culture are performed by routine protocol.

On day 3, each embryo was washed and cultured in single droplets. TE biopsy was conducted and 10μl SCM of biopsied embryos are collected on day 5 or day 6. Both sample types undergo whole-genome amplification (WGA) using Quanti Flour ONE dsDNA system and DNA analysis by next-generation sequencing (NGS) using NextSeq High output 150 cycles kit.

Comparison of NGS results from trophectoderm (TE) biopsy and SCM is done to identify the sensitivity and specificity of the test.

A sample size of 218 day 5/day 6 embryos will be needed.

ELIGIBILITY:
Inclusion Criteria:

* Assisted Reproductive Treatment with ICSI indication
* Having PGT-A or PGT-SR indication
* Having an agreement to be enrolled into NiPGT-A study
* Having blastocyst to biopsy

Exclusion Criteria:

* In vitro maturation cycle

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergo in vitro fertilization.
Sampling Method: Probability Sample
Enrollment: 218 (Estimated)
Dates: Start 2020-08-15 (Actual); Primary Completion 2020-10-31 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of NiPGT-A | 4 months after recruiting
  The ability to detect euploid embryo
Specificity of NiPGT-A | 4 months after recruiting
  The ability to detect aneuploid embryo

SECONDARY OUTCOMES:
Successful amplification rate | 7 days after SCM collection
  Rate of SCM samples with DNA concentration after WGA greater than or equal 1ng/μl
Total concordance | 14 days after SCM collection
  The match NGS results from TE biopsy and SCM for ploidy and sex
Positive pregnancy rate | at 2 weeks after embryo transfer
  Rate of participants with serum human chorionic gonadotropin level greater than 25 mIU/mL
Clinical pregnancy rate | 5 weeks after embryo transfer
  Rate of participants with at least one gestational sac on ultrasound at 7 weeks' gestation with the detection of heart beat activity.
Ongoing pregnancy rate | At 12 weeks' gestation
  Rate of participants with detectable heart at 12 weeks' gestation or beyond, after the completion of the first transfer
Implantation rate | 3 weeks after embryo transfer
  as the number of gestational sacs per number of embryos transferred

CONTACTS AND LOCATIONS:
Overall Officials: Lan N Vuong, Principal Investigator — Mỹ Đức Hospital
Locations (2):
- Vietnam (2):
  - My Duc Phu Nhuan Hospital, Ho Chi Minh City, Phu Nhuan
  - My Duc Hospital, Ho Chi Minh City